CLINICAL TRIAL: NCT00474344
Title: Genetic Linkage Study of Idiopathic Talipes Equinovarus (ITEV) (Clubfoot)
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Other Study IDs: H04-70319
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2017-05

CONDITIONS: Clubfoot
Keywords: Genetics; Clubfoot; DNA; Idiopathic Talipes Equinovarus also known as Clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to identify and characterize the genetic loci causing idiopathic talipes equinovarus (clubfoot).

The hypothesis is that a few genes account for a substantial fraction of ITEV and that these genes can be identified in defined populations. Towards this goal, in preliminary studies, Dr. Hecht's group has identified two genes, NAT2 and CASP10, which demonstrate evidence for linkage and association to ITEV.

DETAILED DESCRIPTION:
Blood Collection: For this study, the investigators need to obtain blood samples from members of families in which clubfoot has occurred; more specifically, blood samples from the affected child and both parents. DNA will be extracted from blood samples. The DNA will then be tested to look for genetic factors that cause clubfoot.

Study Questionnaires: As well as the blood samples, the investigators have a short questionnaire for the mother of the child with clubfoot to complete.

ELIGIBILITY:
Inclusion Criteria:

* One family member, usually child, must have clubfoot

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One family member, usually child, must have clubfoot.
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2004-08; Primary Completion 2010-12 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, Principal Investigator — University of British Columbia
Locations (2):
- University of Texas, Houston, Texas, United States
- BC Children's Hospital, Vancouver, British Columbia, Canada